CLINICAL TRIAL: NCT06319248
Title: MID-STEP (MIDodrine for Sepsis Treatment and Early vasoPressor Weaning) Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ognjen Gajic, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-000121
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Sepsis; Low Blood Pressure
Keywords: Vasopressors
MeSH Terms: conditions — Sepsis; Hypotension | interventions — Midodrine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care Group (Active Comparator)
  Interventions: Other: Standard of Care
- Standard of Care with Midodrine Group (Experimental)
  Interventions: Drug: Midodrine

INTERVENTIONS:
Drug: Midodrine — Subjects will receive standard of care for sepsis and 10 mg of Midodrine every 8 hours administered orally or enterally (via nasogastric tube)
  Arms: Standard of Care with Midodrine Group
Other: Standard of Care — Subjects will receive standard of care for sepsis treatment.
  Arms: Standard of Care Group

SUMMARY:
This study is being done to determine if early administration of Midodrine can improve outcomes by maintaining a higher mean blood pressure off of intravenous medications. Researchers want to see if Midodrine can help people with sepsis need fewer vasopressors, which could mean shorter hospital stays, less time with uncomfortable tubes, and a smoother recovery overall.

ELIGIBILITY:
Inclusion criteria:

Patients diagnosed with sepsis within 24 hours of meeting all of the following criteria will be eligible to participate in the study:

* Sepsis-3 criteria: acute hospital admission for suspected infection with new or worsening organ dysfunction measured by the increase in Sequential Organ failure Assessment (SOFA) score of 2 points or more.
* IV vasopressor use or persistent hypotension (MAP < 65 mm Hg) after initial fluid resuscitation in the ED or ICU (30 mL/kg unless deemed excessive by the treating clinician).

Exclusion criteria:

* High-dose vasopressors (norepinephrine equivalent > 0.3 µg/kg/min).
* Inadequately controlled source of infection.
* Cardiogenic or obstructive (massive pulmonary embolism) shock.
* Clinical suspicion or confirmed diagnosis of bowel obstruction, bowel ischemia, or ileus.
* Contraindication to enteral intake (ileus, vomiting, gastrointestinal bleeding, endoscopic procedures etc.).
* Recent myocardial infarction (within the past 3 months).
* Recent treatment for peripheral vascular disease (within the past 3 months).
* Current use of monoamine oxidase inhibitors.
* Recent stroke (within the past 3 months).
* Prior use of midodrine as a home medication.
* Known allergy to midodrine.
* Comfort care measures.
* Pregnancy.
* Fludrocortisone acetate as a current home medication.
* Bradycardia (heart rate < 50 beats/min).
* Untreated pheochromocytoma.
* Untreated thyrotoxicosis.
* Open-angle glaucoma.
* Treating emergency or critical care physician unwilling to enroll patient in trial.
* Inability to give consent for participation and no representative or surrogate available to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2029-05-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Time alive and without vasopressor support | 28 days
  Measured in hours

SECONDARY OUTCOMES:
Total vasopressor requirements | 28 days
  Measured as norepinephrine equivalents (µg)
Central venous access duration | 28 days
  Measured in hours
Cumulative fluid balance over the first 48 hours | 48 hours
Cumulative fluid balance up to 7 days of ICU stay | 7 days
ICU Length of Stay | 28 days
  Total number of days admitted to the Intensive Care Unit (ICU)
Hospital Length of Stay | 28 days
  Total number of days admitted to the hospital
ICU, hospital, and organ support-free days | 28 days
  Number of ICU, hospital, and organ support-free days

CONTACTS AND LOCATIONS:
Overall Officials: Amos Lal, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No